CLINICAL TRIAL: NCT01113762
Title: Metal-metal Articulations vs Standard 28 mm Cementless Total Hip Arthroplasty in Younger Patients. Randomized Studies
Brief Title: Metal-metal Articulations Versus Standard 28 mm Cementless Total Hip Arthroplasty
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government); Region Zealand (Other); Zimmer Biomet (Industry); DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, jeannette ostergaard penny, MD, PhD, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VF20050133
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Osteoarthritis, Hip
Keywords: Arthroplasty, Replacement, Hip; Bone Density; Rehabilitation; T-Lymphocytes; Chromium Alloys
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- resurfacing (Experimental): a hip replacement that leaves most of the underlying bone intact and mimics the natural biomechanical features of the hip joint
  Interventions: Device: articular surface replacement ASR, DePuy
- large head THA (Experimental): a standard stemmed THA but with a large metal head, and a metal-metal articulation
  Interventions: Device: ReCap/Magnum modular head, Biomet
- 28 mm ceramics-polyethylene (Active Comparator): a standard 28 mm head uncemented THA
  Interventions: Device: Bimetric stem, mallory/head cup, 28 mm ceramic head, Biomet
- 28 mm metal-polyethylene THA (Active Comparator): a standard stemmed uncemented THA
  Interventions: Device: 28 mm CrCo head, Trilogy CH cup, VerSys Fiber stem,Zimmer)

INTERVENTIONS:
Device: articular surface replacement ASR, DePuy — posterolateral incision
  Arms: resurfacing
Device: ReCap/Magnum modular head, Biomet — posterolateral incision
  Arms: large head THA
Device: Bimetric stem, mallory/head cup, 28 mm ceramic head, Biomet — posterolateral incision
  Arms: 28 mm ceramics-polyethylene
Device: 28 mm CrCo head, Trilogy CH cup, VerSys Fiber stem,Zimmer) — posterolateral incision
  Arms: 28 mm metal-polyethylene THA

SUMMARY:
Younger hip patients often need revision of their hip replacement due to wear and loosening. Newer concepts (resurfacing and large head total hip replacement) with articulation surfaces in metal may reduce the wear, increase the longevity of the implant and give an improved function. The possible downside is that these concepts releases metal debris to the body. The investigators wish to see if the newer interventions are a clinical improvement compared to standard. The investigators also wish to investigate the extent of metal released to the body and any effect on the immune system. Finally the investigators wish to investigate the stability of these new implants and their ability to preserve the bone around the implant.

The investigators hypothesis is:

That the metal on metal articulations will not have better clinical outcomes than standard The resurfacing implant is expected to preserve the bone of the upper femoral bone. The implants are expected to be stabile within the first year.

ELIGIBILITY:
Inclusion Criteria:

* Primary hip osteoarthritis
* Secondary osteoarthritis due to mild dysplasia
* Age from 40 to 65 years

Exclusion Criteria:

* Dysplasia with CE angle < 25 degrees on the AP projection
* Severe femoral head deformation
* Reduced femoral neck length
* Leg length discrepancy more than 1 cm
* Need for restoration of offset
* Deformation after fractures or earlier osteotomies
* A previous hip arthroplasty
* Inflammatory arthritis
* Endocrinological disease with bone metabolic manifestations
* Renal disease
* Malignant disease
* Neuro/muscular or vascular diseases of the affected leg
* Osteoporosis
* Use of opioid pain killers due to other diseases
* High dose corticosteroids
* Obese with BMI > 35
* Pregnant or planning to be
* Ppresented problems that would prevent completing our follow-up program

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2007-02; Primary Completion 2009-11 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Range of motion | Up to two months before surgery
  range of motion in the hip joint evaluated by goniometer
Range of motion | 8 weeks +/- 1 week
  Range of motion of the hip joint
Range of motion | 6 months +/- 2 weeks
  range of motion in the hip joint
Range of motion | 1 year +/- 1 month
  range of motion in the hip joint
range of motion | 2 year +/- 1 month
  range of motion in the hip joint

SECONDARY OUTCOMES:
Metal ions | Up to two months before surgery
  Crome and cobalt ions in serum and whole blood.
BMD | Within the first week following surgery
  bone mass density around the implants
RSA | Within the first week following surgery
  radiostereommetry. Measurement of micromotions (subsidence, rotation and translations)of the implant in relation to the bone
HHS | Up to two months before surgery
  Harris hip score. An investigator asssesed hip questionnaire including pain, function, deformities and range of motion
UCLA activity | Up to two months before surgery
  University of California Los Angeles activity score. A score over the intensity of activities the patient engages in.
WOMAC | Up to two months before surgery
  patient reported outcome of pain, stifness and disability during activities of daily living.
EQ-5d | Up to two months before surgery
  a short quality of life measure. patient reported
T cell count | Up to two months before surgery
  quantitative analysis of the level of T-cells in the blood
X-ray | within 2 years of surgery
  an assesment of the placement of the metal cup. Inclination and anteversion.
steps | Up to two months before surgery
  using a pedometer 1 week prior to each check up the annual step rate is calculated
sick leave | assesed 6 months following surgery.
  an assesment of the rehabilitation period following the intervention
Metal ions | 8 weeks +/- 1 week
  Crom and cobalt
Metal ions | 6 months +/- 2 weeks
  Crome and cobalt
Metal ions | 1 year +/- 1 month
  crome and cobalt
metal ions | 2 year +/- 1 month
  crome and cobalt
BMD | 8 weeks +/- 1 week
  bone mass desity around the implant
BMD | 1 year +/- 1 month
  Bone mass density around the implant
BMD | 2 year +/- 1 month
  Bone mass density around the implant
RSA | 8 weeks +/- 1 week
  Radiostereometry of implant
RSA | 6 months +/- 2 weeks
  Radiostereometry of implant
RSA | 1 year +/- 1 month
  Radiostereometry of implant
RSA | 2 year +/- 1 month
  Radiostereometry of implant
HHS | 8 weeks +/- 1 week
  Harris hip score
HHS | 6 months +/- 2 weeks
  Harris hip score
HHS | 1 year +/- 1 month
  Harris hip score
HHS | 2 years +/- 1 month
  Harris hip score
UCLA activity | 8 weeks +/- 1 week
  activity score
UCLA activity | 6 months +/- 2 weeks
  activity score
UCLA activity | 1 year +/- 1 month
  activity score
UCLA activity | 2 years +/- 1 month
  activity score
WOMAC | 3 weeks
  self reported function
WOMAC | 6 weeks
  self reported function
WOMAC | 8 weeks +/- 1 week
  self reported function
WOMAC | 6 months +/- 2 weeks
  self reported function
WOMAC | 1 year +/- 1 month
  self reported function
WOMAC | 2 years +/- 1 month
  self reported function
EQ-5d | 8 weeks +/- 1 week
  quality of life
EQ-5d | 6 months +/- 2 weeks
  quality of life
EQ-5d | 1 year +/- 1 month
  quality of life
EQ-5d | 2 years +/- 1 month
  quality of life
T cell count | 8 weeks +/- 1 week
  T cell count
T cell count | 6 months +/- 2 weeks
  T cell count
T cell count | 1 year +/- 1 month
  T cell count
T cell count | 2 years +/- 1 month
  T cell count
steps | 8 weeks +/- 1 week
  steps measured by pedometer during the week prior to check up
steps | 6 months +/- 2 weeks
  steps measured by pedometer during the week prior to check up
steps | 1 year +/- 1 month
  steps measured by pedometer during the week prior to check up
steps | 2 years +/- 1 month
  steps measured by pedometer during the week prior to check up
blood loss | during surgery
  blood loss measured in mL
days in hospital | from admission to discharge from hospital
  days in hospital following surgery
complications | within the first 2 years following surgery
  surgery and implant related complications
surgery time | during surgery
  time from skin is incised to skin is closed
incision length | during surgery
  the length of the surgical incision in cm

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Overgaard, MD, professor, phd, Principal Investigator — University of Southern Denmark
Locations (2):
- Denmark (2):
  - Naestved Hospital Dept. of orthop. surg., Næstved
  - Odense University hospital, Odense

REFERENCES:
- [Derived] Penny JO, Varmarken JE, Ovesen O, Nielsen C, Overgaard S. Metal ion levels and lymphocyte counts: ASR hip resurfacing prosthesis vs. standard THA: 2-year results from a randomized study. Acta Orthop. 2013 Apr;84(2):130-7. doi: 10.3109/17453674.2013.784657. PMID 23597114
- [Derived] Penny JO, Ovesen O, Varmarken JE, Overgaard S. Similar range of motion and function after resurfacing large-head or standard total hip arthroplasty. Acta Orthop. 2013 Jun;84(3):246-53. doi: 10.3109/17453674.2013.788435. Epub 2013 Mar 26. PMID 23530872
- [Derived] Nissen T, Douw K, Overgaard S. Patient-reported outcome of hip resurfacing arthroplasty and standard total hip replacement after short-term follow-up. Dan Med Bull. 2011 Oct;58(10):A4310. PMID 21975150